CLINICAL TRIAL: NCT01802242
Title: Tumor Targeted Radiotherapy for Patients With Localized Prostate Cancer
Brief Title: Tumor TARGET Prostate Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB 12-5015-C
Record Dates: First submitted 2012-10-22; First posted 2013-03-01 (Estimated); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Prostate tumour; Prostate radiotherapy; prostate cancer treatment
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy, Intensity-Modulated; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Radiation Treatment (Cohort 2) (Experimental)
  Interventions: Radiation: Volumetric Modulated Arc Therapy (VMAT) and High-Dose Rate (HDR) Radiotherapy
- Prior Radiation Treatment (Control Cohort) (Other): Patients who received 78Gy RT to the prostate gland 3-4.5 years prior to enrollment. This group will not be receiving any active treatment
  Interventions: Other: No Active Treatment - completed Prior Radiation

INTERVENTIONS:
Radiation: Volumetric Modulated Arc Therapy (VMAT) and High-Dose Rate (HDR) Radiotherapy — Patients in this group will receive one of 2 treatment arms of their choice:
  * Arm 1: VMAT delivery with integrated VMAT boost (IB-VMAT) GTV: 95Gy in 38fractions
  * Arm 2: HDR-boost followed by VMAT GTV: 10Gy HDR + 76Gy in 38 fractions VMAT
  Arms: Active Radiation Treatment (Cohort 2)
Other: No Active Treatment - completed Prior Radiation — Already had prior radiation treatment. MRI-guided prostate biopsy at 3 years and PSA per standard practice
  Arms: Prior Radiation Treatment (Control Cohort)

SUMMARY:
Prostate cancer is common in males and may develop over the course of an individual's life. This cancer is often discovered at the time of routine physical examinations and/or blood work or on rectal examination. Once diagnosed, most patients do require some form of treatment so that the prostate cancer does not progress to cause damage and/or shortened lifespan. Occasionally, after patients receive treatment, the investigators have found that an area of cancer remains within the prostate. Those patients with a large area of cancer (i.e. seen on MRI image) appear to have a higher chance of remaining or recurrent prostate cancer even after standard treatment. Thus, the investigators believe that the area of the prostate gland occupied by a dense area of cancer may need more radiation therapy than normal to remain cancer free.

Standard therapy currently in place in North America: Currently patients who are diagnosed with prostate cancer have 3 common options: surgery, external beam radiation therapy (EBRT) alone or internal radiation (brachytherapy). Patients may or may not receive hormone therapy alongside the radiation depending on their physician's preference. For those who receive radiation therapy, the tumor typically receives the same dose as the rest of the prostate gland.

Findings to date: In the past few years the investigators have discovered that patients with a tumor large enough to be seen on MRI images (>5mm) have a higher chance than normal of having cancer remain in the prostate, despite receiving treatment for their cancer 3 years earlier. Using new technology investigators can deliver radiation therapy after viewing the prostate tumor on MRI. This guides therapy, allowing the radiation treatment to be targeted to the tumor within the prostate. Based on this earlier success the investigators believe that they can now safely give a higher dose of radiation to specifically target the cancer within the prostate gland.

Reason for the study: The investigators would like to test this technology and expertise to give radiation to a higher than normal dose to the tumor nodule in prostate gland.

DETAILED DESCRIPTION:
This is a prospective two arm phase 2 trial investigating the technical and clinical performance of tumor-targeted (rather than prostate targeted) radiotherapy.

Cohort 1 (Control group): This group consists of patients who have had previous radiation. This group will not receive any active treatment but will have a biopsy at 3 years from the time they completed their radiation therapy. Patient in this group will also continue to have their PSA checked per standard practice

Cohort 2 (Experimental group): Patients in this group will receive one of 2 treatment arms of their choice. In addition to the MRI-guided prostate biopsy at 3 years and regular standard of care PSA checks, this group will also complete a quality of life questionnaire and have regular imaging per standard practice.

Both groups will be followed by the research team per protocol.

ELIGIBILITY:
Inclusion Criteria [applicable to both Cohorts 1 (control) and Cohort 2 (Experimental) unless otherwise specified]:

1. Histological evidence of prostate adenocarcinoma.
2. Discrete intra-prostatic tumor that can be confidently visualized on MRI prior to radiotherapy (>5mm maximum diameter but <33% of prostate volume, biopsy confirmed from initial diagnosis or interventional Biopsy) )
3. At least 18 years old
4. ECOG performance status 0 or 1 with > 10-year life expectancy
5. Informed consent: All patients must sign a document of informed consent indicating their understanding of the investigational nature and risks of the study before any protocol related studies are performed (this does not include standard care laboratory tests or imaging studies).
6. Patients will be one of the following risk groups prior to therapy:

   * Low-risk disease (Gleason 6 and PSA <10 and T1) AND >50% of biopsy cores involved with tumor
   * Intermediate-risk disease (Gleason 7 or PSA 10-20 or T2)
   * High-risk disease (Gleason >8 or T3 or PSA >20)
7. Risk of LN involvement <30% (Roach formula = 2/3PSA([G-6]x10))
8. Patients who received 78Gy RT to the prostate gland 3-4.5 years prior to enrollment (Cohort 1 only)

Exclusion Criteria [applicable to both Cohorts 1 (control) and Cohort 2(Experimental) unless otherwise specified]:

1. Previous history of radiation therapy to the prostate (Cohort 2)
2. Diagnosis of another cancer not being skin cancer within the last 5 years (Cohort 2)
3. Patients weighing >136kgs (weight limit for the scanner tables)
4. Patients with contraindications to MRI: this includes patients with pacemakers, cerebral aneurysm clips, shrapnel injury or implantable electronic devices not compatible with MRI determination. Exceptions will be allowed if deemed sage and appropriate by the MRI technologist.
5. Severe claustrophobia
6. Bleeding diathesis and anti-coagulative therapy that cannot be temporarily ceased precluding biopsy
7. Current hormonal therapy (Cohort 1) or initiated >2 weeks prior to enrollment (Cohort 2)
8. Radiological evidence of regional or distant metastases (Cohort 2)
9. Other urinary or medical conditions deemed by the PI or associates to make the patient ineligible for MRI-guided prostate biopsy
10. Contraindications to the endorectal coil, surgically absent rectum, severe hemorrhoids or previous colorectal surgery
11. Contraindications to conscious sedation
12. Latex allergy
13. History of Ulcerative Colitis, Crohn's Disease, Ataxia Telangiectasia, or SLE (Cohort 2)
14. Other medical conditions deemed by the PI to make patient ineligible for study intervention

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2012-10; Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Determine rates of Local Control after standard targeted boost radiotherapy in patients with localized prostate cancer. | 5 years

SECONDARY OUTCOMES:
Determine if high-dose tumor-targeted radiotherapy for localized prostate cancer can be integrated in a standard-care workflow. | 5 years
Determine a methodology with appropriate uncertainty margins for Gross Tumour Volume boost | 5 years
Evaluate the spatial distribution of prostatic carcinoma at the time of repeat biopsy | 5 years
Compare dose to recurrent and non-recurrent tumor nodules. | 5 years
Determine rates of toxicity with tumor-targeted boost radiotherapy. | 5 years
Assess Quality of Life (QoL) outcomes after high-dose tumor-targeted boost therapy. | 5 years
Determine patient acceptance of combination of high dose rate and volumetric modulated arc therapy techniques | 5 years
Determine clinical outcomes by comparing integrated boost volumetric modulated arc therapy and a combination of high dose rate and volumetric modulated arc therapy techniques. | 5 years
Determine dosimetric outcomes by comparing integrated boost volumetric modulated arc therapy and a combination of high dose rate and volumetric modulated arc therapy techniques. | 5 years

OTHER OUTCOMES:
Explore the predictive value of baseline and early response imaging biomarkers on Local Control. | 5 years
Bank tissue and biofluids for future exploration of the relationship between biopsy tissue/serum/urine and disease recurrence. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter Chung, MB ChB, Principal Investigator — University Health Network, The Princess Margaret
Locations (1):
- University Health Network, The Princess Margaret, Toronto, Ontario, Canada